CLINICAL TRIAL: NCT02357862
Title: Impact of Mitral Valve Annuloplasty on the Tricuspid Valve Complex
Brief Title: Changes in the Tricuspid Valve Complex Induced by Mitral Valve Annuloplasty
Status: Terminated | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: MVR_TV
Record Dates: First submitted 2015-01-26; First posted 2015-02-06 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2015-07

CONDITIONS: Tricuspid (Valve); Deformity
Keywords: Cardiovascular Diseases; Heart Valve Diseases; Mitral Valve Annuloplasty; Tricuspid Valve Insufficiency
MeSH Terms: conditions — Congenital Abnormalities; Cardiovascular Diseases; Heart Valve Diseases; Tricuspid Valve Insufficiency | interventions — Mitral Valve Annuloplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mitral Valve Annuloplasty: All eligible patients
  Interventions: Procedure: Mitral Valve Annuloplasty

INTERVENTIONS:
Procedure: Mitral Valve Annuloplasty — Mitral valve annuloplasty by a rigid mitral ring, a semi-rigid ring, or a fully flexible band, at the surgeon's discretion

SUMMARY:
The purpose of this study is to evaluate the impact of isolated mitral valve annuloplasty on the geometry and the function of the tricuspid valve complex.

DETAILED DESCRIPTION:
The proposed pathogenesis of functional tricuspid regurgitation (TR) in mitral valve disease seems incomplete. Because both atrioventricular valves are closely connected to each other by means of the cardiac fibrous skeleton, the geometry of the tricuspid valve is likely to be distorted after ring-annuloplasty of the mitral valve. This could lead to the development of functional TR, or to an increase in TR severity. To test this hypothesis, a prospective study will be started in patients undergoing isolated mitral valve annuloplasty.

ELIGIBILITY:
Inclusion Criteria:

* all patients 18 years of age or older undergoing minimally invasive, isolated mitral valve annuloplasty

Exclusion Criteria:

* concomitant tricuspid valve surgery
* atrial fibrillation at the moment of surgery
* poor echocardiographic windows

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing minimally invasive, isolated mitral valve annuloplasty in the University Hospitals Leuven
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Postoperative geometric changes in tricuspid valve annulus (TA) | day 0
  Measurement of changes in 3D descriptors of the TA (e.g. changes from baseline in the TA area of the best-fit plane in cm^2, and changes from baseline in the height of each TA point to the TA best-fit plane in mm)

CONTACTS AND LOCATIONS:
Overall Officials: Werner Budts, M.D., PhD, Principal Investigator — KU Leuven - University of Leuven, Department of Cardiovascular Sciences, Division of Cardiology; University Hospitals Leuven, Department of Cardiology